CLINICAL TRIAL: NCT04035317
Title: Effect of Aesculus Hippocastanum L. (Sapindaceae, "Horse Chestnut") on Fontan Circulation - a Randomized Clinical Trial
Brief Title: Aesculus Hippocastanum L. on Fontan Circulation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The graduate student quit.
Sponsor: Casa Espirita Terra de Ismael (Other)
Collaborators: Hospital das Clínicas de Ribeirão Preto (Other)
Responsible Party: Principal Investigator, Fabio Carmona, MD, PhD, Casa Espirita Terra de Ismael
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CastanhaFontan
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Univentricular Heart
Keywords: Fontan operation; Aesculus hippocastanum; mesenteric artery resistance
MeSH Terms: conditions — Univentricular Heart | interventions — horse chestnut seed

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive Aesculus hippocastanum or placebo for 4 months, followed by 4 weeks of washout and crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The capsules will be identical in appearance and will be labelled only with patient's name.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aesculus hippocastanum (Experimental): Patients will receive extract of Aesculus hippocastanum
  Interventions: Drug: Aesculus Hippocastanum / Horse Chestnut
- Placebo (Placebo Comparator): Patients will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aesculus Hippocastanum / Horse Chestnut — Treatment for 4 months, washout of 4 weeks, then crossover for another 4 months.
  Arms: Aesculus hippocastanum
Drug: Placebo — Treatment for 4 months, washout of 4 weeks, then crossover for another 4 months.
  Arms: Placebo

SUMMARY:
Patients after the Fontan operation at a single institution will be randomized to receive a standardized extract of Aesculus hippocastanum L. (horse chestnut) or placebo for 4 months in a crossover clinical trial. The primary outcome will be the mesenteric artery resistance measured by Dopple sonography.

ELIGIBILITY:
Inclusion Criteria:

* Underwent Fontan surgery

Exclusion Criteria:

* Severe adverse reaction
* Personal or parental request

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mesenteric artery resistance | After 4 months
  Mesenteric artery resistance, measured by pulsed-wave Doppler, in 0.1 units

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil